CLINICAL TRIAL: NCT05141617
Title: Endoscopic Treatment vs Transjugular Intrahepatic Portosystemic Shunt in the Management of Oxaliplatin Related Gastroesophageal Variceal Bleeding: A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Management of Oxaliplatin-related Gastroesophageal Variceal Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Shanghai Minhang Central Hospital (Other); Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLAEGV-TRE
Record Dates: First submitted 2021-11-01; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Gastroesophageal Varices Hemorrhage; Gastrointestinal Cancer; Received Oxaliplatin-based Chemotherapy
Keywords: portal hypertension; Gastrointestinal Cancer; oxaliplatin; gastroesophageal variceal bleeding; endoscopic treatment; Transjugular Intrahepatic Portosystemic Shunt
MeSH Terms: conditions — Gastrointestinal Neoplasms; Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic treatment group (Experimental): Patients in the endoscopic treatment group receive endoscopic variceal ligation and N-butyl-cyanoacrylate according to the type of varices.
  Interventions: Procedure: Endoscopic treatment
- TIPS group (Experimental): Patients in the TIPS group receive transjugular intrahepatic portosystem stent-shunt.
  Interventions: Procedure: TIPS

INTERVENTIONS:
Procedure: Endoscopic treatment — Patients in the endoscopic treatment receive endoscopic variceal ligation and N-butyl-cyanoacrylate according to the type of varices
  Arms: Endoscopic treatment group
Procedure: TIPS — Patients in the TIPS group receive Transjugular Intrahepatic Portosystemic Shunt
  Arms: TIPS group

SUMMARY:
In this randomized controlled study, we aim to compare the efficacy and safety of these two interventions in patients with oxaliplatin-induced gastroesophageal variceal bleeding.

DETAILED DESCRIPTION:
Oxaliplatin is used as the first-line chemotherapy for colorectal cancer. However, oxaliplatin-induced hepatotoxicity could lead to sinusoidal injury and portal hypertension in the long term. Variceal bleeding, as the most common complication of portal hypertension, threaten these patents' life. Endoscopic treatment and Transjugular Intrahepatic Portosystemic Shunt (TIPS) are both recommended management of gastroesophageal variceal bleeding. In this randomized controlled study, we aim to compare the efficacy and safety of these two interventions in patients with oxaliplatin-induced gastroesophageal variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Having received oxaliplatin-based chemotherapy for at least one cycle
2. History of variceal bleeding (including hematemesis or melena)
3. Portal hypertension confirmed by CT or MRI
4. Esophageal and / or gastric varices confirmed by endoscopy
5. Informed consent signed

Exclusion Criteria:

1. With serious life-threatening diseases of circulation / blood / respiratory system
2. With known causes of liver cirrhosis (hepatitis B, hepatitis C, autoimmune, schistosomiasis, non-alcoholic fatty liver disease, and etc.)
3. With contraindications of endoscopic treatments and TIPS;
4. Participation refused

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
24-week re-bleeding | 24 weeks
  Hematemesis ,melena, or hemoglobin level decreased by 10 g/L within 6 hours

SECONDARY OUTCOMES:
8-week re-bleeding | 8 weeks
  Hematemesis ,melena, or hemoglobin level decreased by 10 g/L within 6 hours
8-week mortality | 8 weeks
  death
8-week adverse events | 8 weeks
  Other complications of portal hypertension such as the progression of ascites, liver failure, etc.
24-week mortality | 24 weeks
  death
24-week adverse events | 24 weeks
  Other complications of portal hypertension such as the progression of ascites, liver failure, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao CHENCHEN, M.D. & Ph.D, Principal Investigator — Fudan University
Locations (1):
- Department of Gastroenterology and Hepatology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Huang X, Li F, Wang L, Xiao M, Ni L, Jiang S, Ji Y, Zhang C, Zhang W, Wang J, Chen S. Endoscopic treatment of gastroesophageal variceal bleeding after oxaliplatin-based chemotherapy in patients with colorectal cancer. Endoscopy. 2020 Sep;52(9):727-735. doi: 10.1055/a-1157-8611. Epub 2020 May 7. PMID 32380558